CLINICAL TRIAL: NCT02922348
Title: Optimal Hormone Replacement for Women With Premature Ovarian Insufficiency
Brief Title: Hormone Replacement for Premature Ovarian Insufficiency
Acronym: HOPE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 823553
Record Dates: First submitted 2016-03-21; First posted 2016-10-04 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Primary Ovarian Insufficiency
Keywords: premature ovarian failure; hormone replacement
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Hormone Replacement Therapy; Estradiol; Progesterone; Medroxyprogesterone; Medroxyprogesterone Acetate; Contraceptives, Oral, Combined; Ethinyl Estradiol; norgestimate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hormone Replacement Therapy (Experimental): Patient will be given hormones in the form of: transdermal estradiol patch (Climara) 100 mcg/24 hours weekly, progesterone (Prometrium) 200 mg per day for first 12 calendar days of each month (If patients insurance plan does not cover transdermal estradiol, they will be prescribed oral estradiol 2 mg daily. If patients insurance plan does not cover Prometrium, they will be prescribed medroxyprogesterone (Provera) 10 mg per day for first 12 calendar days of each month).
  Interventions: Drug: Hormone Replacement Therapy
- Combined Oral Contraceptives (Experimental): Patients will be given hormones in the form of: monophasic combined oral contraceptive containing ethinyl estradiol 0.035 mg and norgestimate 0.25 mg, 1 tablet daily (21 days of active pills and 7 days of inactive pills)
  Interventions: Drug: Combined Oral Contraceptives

INTERVENTIONS:
Drug: Hormone Replacement Therapy — Hormone replacement therapy as indicated in Arm 1
  Other Names: Estradiol; Prometrium; Micronized progestin; Medroxyprogesterone; Climera; Provera
  Arms: Hormone Replacement Therapy
Drug: Combined Oral Contraceptives — Combined oral contraceptives as indicated in Arm 2
  Other Names: Ethinyl estradiol; Norgestimate
  Arms: Combined Oral Contraceptives

SUMMARY:
The investigators intend to establish feasibility/acceptability of a pilot randomized trial comparing hormone replacement therapy (HRT) and combined oral contraceptives (COCs) in women with premature ovarian insufficiency to estimate differences in quality of life (QOL) and serum hormone assays and markers of bone turnover/cardiovascular risk. At baseline, QOL survey will be administered and serum testing performed. Patients then randomized to HRT or COCs. Repeat testing will be performed after 3 and 6 months.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) is a term used to describe when a woman's ovaries stop working normally before the natural age of menopause. Early sequelae of POI include vasomotor symptoms, vaginal dryness, mood swings and insomnia due to estrogen deficiency. Long-term sequelae such as loss of bone mineral density and cardiovascular risk carry are considerable concerns. While exogenous estrogen replacement is recommended for the POI patient population, the optimal regimen for replacement is not clear. One approach to hormone replacement therapy (HRT) is to mimic physiologic ovarian function through full replacement doses of estrogen (either orally or transdermally) to reach the typical serum estradiol levels of a menstruating woman (approximately 104 pg/mL per day) with cyclic progestin therapy for endometrial protection. Another approach uses daily combined estrogen-progestin oral contraceptives (COCs), for ease of administration and increased social acceptability. To date, few studies have been performed comparing the two treatment methods in terms of quality of life measures (vasomotor symptoms, bleeding profile, sexual dysfunction, satisfaction with contraception), endocrine function, bone turnover or cardiovascular risk in POI patients. In this proposal, the investigators intend to establish feasibility and acceptability of a pilot randomized controlled trial comparing traditional HRT with COCs in women with POI and to evaluate differences in quality of life measures, hormone assays, bone turnover and cardiovascular risk between treatment arms. The investigators hypothesize that acceptability and feasibility of the pilot trial will be high and that differences will be detected for all measured variables between treatment arms. Demonstration of feasibility and acceptability of this pilot would allow for the pursuit of a larger trial and identification of a superior treatment regimen would have a meaningful impact on the short and long-term care of this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Female patients,
* Between 14-45 years of age
* Post-menarchal
* Presence of uterus
* POI as defined by: change in menstrual function (oligomenorrhea and/or amenorrhea), elevated serum serum follicle stimulating hormone (FSH), low serum estradiol concentrations, or estrogen deficiency symptoms.

Exclusion Criteria:

* Pregnancy or lactation within previous 3 months
* Use of hormonal contraception or replacement within previous 3 months
* Any contraindication to oral contraceptive pills or hormone replacement therapy per the current drug labels. These could include, but are not limited to: history of venous thromboembolism,estrogen-sensitive cancer history, regular cigarette smoking and history of or active liver disease, etc.
* Patients will be screened for pregnancy with a urine HCG test at time of screening

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | 1 year
  Patient willingness to participate and be randomized

SECONDARY OUTCOMES:
Vasomotor symptoms - Greene Climacteric Scale | 1 year
  Greene Climacteric Scale
Vasomotor symptoms - Menopausal Vasomotor Symptoms (MVS) survey | 1 year
  Menopausal Vasomotor Symptoms (MVS) survey
Bleeding profile - Bleeding questionnaire | 1 year
  Bleeding questionnaire
Bleeding profile - Menstrual diary | 1 year
  Menstrual diary
Sexual dysfunction - Female Sexual Function Index (FSFI) | 1 year
  Female Sexual Function Index (FSFI)
Satisfaction as Contraceptive Method | 1 year
  Birth Control Satisfaction Assessment
Hormone Assays - FSH (mIU/mL) | 1 year
  FSH (mIU/mL)
Hormone Assays - Estradiol (pg/mL) | 1 year
  Estradiol (pg/mL)
Hormone Assays - Sex-hormone binding globulin (nmol/L) | 1 year
  Sex-hormone binding globulin (nmol/L)
Hormone Assays - Total testosterone (ng/dL) | 1 year
  Total testosterone (ng/dL)
Hormone Assays - Free testosterone (ng/dL) | 1 year
  Free testosterone (ng/dL)
Hormone Assays - Anti-mullerian hormone (pmol/l) | 1 year
  Anti-mullerian hormone (pmol/l)
Hormone Assays - Dehydroepiandrosterone Sulfate (ng/mL) | 1 year
  Dehydroepiandrosterone Sulfate (ng/mL)
Hormone Assays - Thyroid stimulating hormone (U/mL) | 1 year
  Thyroid stimulating hormone (U/mL)
Bone Turnover Markers - Serum osteocalcin (ng/mL) | 1 year
  Serum osteocalcin (ng/mL)
Bone Turnover Markers - Serum N-telopeptide of type I collagen (nmol/L) | 1 year
  Serum N-telopeptide of type I collagen (nmol/L)
Cardiovascular Risk Markers - Total cholesterol | 1 year
  Total cholesterol (mg/dL)
Cardiovascular Risk Markers - Triglycerides (mg/dL) | 1 year
  Triglycerides (mg/dL)
Cardiovascular Risk Markers - Lipoprotein a (mg/dL) | 1 year
  Lipoprotein a (mg/dL)
Cardiovascular Risk Markers - Fasting glucose (mg/dL) | 1 year
  Fasting glucose (mg/dL)
Cardiovascular Risk Markers - Fasting insulin (pmol/L) | 1 year
  Fasting insulin (pmol/L)
Cardiovascular Risk Markers - Homeostatic model assessment (HOMA) insulin | 1 year
  Homeostatic model assessment (HOMA) insulin
Cardiovascular Risk Markers - Tissue-type plasminogen activator antigen (ng/mL) | 1 year
  Tissue-type plasminogen activator antigen (ng/mL)
Cardiovascular Risk Markers - Plasma plasminogen activator inhibitor 1 (ng/mL) | 1 year
  Plasma plasminogen activator inhibitor 1 (ng/mL)
Cardiovascular Risk Markers - Fibrinogen (mg/dL) | 1 year
  Fibrinogen (mg/dL)
Cardiovascular Risk Markers - Factor VII (%) | 1 year
  Factor VII (%)
Cardiovascular Risk Markers - C-reactive protein (mg/L) | 1 year
  C-reactive protein (mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Fertility Care, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No